CLINICAL TRIAL: NCT07078227
Title: 5 Years Follow-up of the Study: "Pharmacogenetics in Depressed Patients With Specific Focus on Difficult-to-treat Depresssion, Suicide Attempt and CYP2D6"
Brief Title: Long-term Follow-up of Depressive Disorders in Psychiatric Care
Status: Not yet recruiting | Type: Observational
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-04820-02
Record Dates: First submitted 2025-03-13; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-06

CONDITIONS: Depression; Psychiatric Diagnosis; Personality Disorders; Suicide, Attempted; CYP2D6 Polymorphism; Anhedonia
MeSH Terms: conditions — Depression; Mental Disorders; Personality Disorders; Suicide, Attempted; Anhedonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention is used. — No intervention is used.

SUMMARY:
The project investigates long-term prognosis and predictors of treatment outcomes for difficult-to-treat depression in patients in secondary psychiatric care. The current patient cohort was collected in 2012-2021 in the study "Pharmacogenetics in patients with depression with specific focus on difficult-to-treat depression, suicide attempt and CYP2D6". The cohort consists of 415 patients, examined carefully regarding diagnostic assessment and earlier treatment. All participants were also genotyped for the drug metabolizing enzymes CYP2D6 and CYP2C19. Blood samples were stored in biobank for other analyses linked to prognostic markers.

The patient cohort will now be followed up with a review of medical records and extraction of register data for a period of 5 years after their participation in the original study. The purpose of the study is to improve treatment and increase knowledge about long-term prognosis in difficult-to-treat depression. This is done by examining symptom profiles, monitoring clinical course and suicidality, and examining prognostic markers.

DETAILED DESCRIPTION:
BACKGROUND

It is very important to understand the course of depressive disorders over time in long time follow-up studies. A cross-sectional observational study "Pharmacogenetics in depressed patients with a special focus on difficult-to-treat depression, suicide attempts and CYP2D6" (n=415) was performed in Sweden 2012-2021. Participants were genotyped for enzymes within the Cytochrome P450 system - CYP2D6 and CYP2C19. Participants were also examined very carefully with regard to diagnostic assessment with structured and semi-structured diagnostic instruments: MINI neuropsychiatric interview (MINI) and structured clinical interview for DSM-IV-TR axis II (SCID-II). Comprehensive psychipatological rating scale (CPRS) was used as well as Montgomery Asberg depression rating scale (MADRS), the UKU side effect rating scale (UKU-SERS) , Suicidal assessment scale (SUAS) and Alcohol Use Disorder Identification Test (AUDIT) and Drug Use Disorder Identification Test (DUDIT) as well as thorough survey of the clinical course of psychiatric symptoms. Blood samples were collected and stored in biobank. The participants with CYP2D6UM and CYP2D6PM were offered pharmacological counseling to optimize treatment during 8 weeks.

The same patients will now be followed over a five-year period after participation in the original study, in order to better understand the long-term prognosis of depression and the factors that can predict the course of the disorder over time.

OBJECTIVE

The overall goal is to improve treatment and increase knowledge about difficult-to-treat depression, as well as to investigate how biological and clinical variables can predict treatment outcomes and long-term outcomes.

PURPOSE

To investigate diagnoses and diagnostic assessment, long-term prognosis, symptom profiles and prognostic markers as well as suicidality and effect of pharmacologic counseling in depression. The cohort contains patients with both unipolar and bipolar depression.

METHOD

Research subjects who have participated in the original study during the period 2012-2021 (n=415) will participate in the follow up study unless they oppose to do so. The original study has already been presented in earlier publications with regard to diagnostics treatment linked to clinical parameters and suicide attempts, inflammation, vitamin D, mitochondrial DNA, CYP2D6, and coping.

Data collection for this follow-up study is based on an approved opt-out procedure from the Swedish Ethical Review Authority (dnr: 2024-04820-02 and 2025-03351-02)). Participants are given the opportunity to decline participation in the study by responding via letter or questionnaire responses digitally. If participants do not respond within 4 weeks, they are automatically included in the study.

Data will be collected through medical records review and extraction of register data. The data collection will be for a period of 5 years from participation in the original study.

The following information is collected from medical records: Information on suicide attempts, inpatient treatment, emergency room visits, outpatient visits, treatment received, ICD diagnoses, descriptions of personality functioning, markers for clinical improvement, if CYP2D6UM and CYP2D6PM have been subject to specific considerations in choice of drug treatment.

Registers will be used when needed for data collection, from the Longitudinal Integration Database for Health Insurance and Labour Market Studies, the Pharmaceutical Register, the Patient Register, the Cause of Death Register.

ELIGIBILITY:
Inclusion Criteria:

Participation in the study "Pharmacogenetics in depressive patients with specific focus on difficult-to-treat depression, suicide attempt and CYP2D6"

Exclusion Criteria:

Not wanting to participate in the follow-up study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 415 patients from the study "Pharmacogenetics in depressive patients with specific focus on difficult-to-treat depression, suicide attempt and CYP2D6". The study population has been well described in earlier publications.
Sampling Method: Non-Probability Sample
Enrollment: 415 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Suicide attempt and suicide | 5 years follow-up after baseline visit.
  The frequency of suicide attempts and completed suicides in the patient sample over the follow-up period of 5 years
Clinical course of depression | 5 years follow-up after baseline visit
  Course of depressive disorder during the follow-up period measured by information from medical records, where the reserach psychiatrist makes an assessment dichotomized as improved or not improved based on the available information.
Comparison of diagnostic assessment for personality disorders | Baseline data and 5 years follow-up from inclusion.
  Comparison of frequency of DSM-IV-TR personality disorders and ICD-11 personality disorders in the sample. ICD-11 personality disorders will also be divided into degree of difficulty as well as which specifiers of prominent traits are present in the population of difficult-to-treat depression
Course and diagnostic characteristics of bipolar disorder | Baseline data and 5 years follow-up after inclusion.
  Historical order of diagnoses before bipolar diagnosis and the development of diagnostic assessment during follow-up as well as personality assessment according to DSM-IV and ICD-11.
Results from pharmacological counseling for CYP2D6UM och CYP2D6PM | Nine weeks of pharmacological counseling after baseline and 5 years follow-up from baseline visit
  Change in score for Montgomery Åsberg Depression Rating Scale from week 0 to 8 (total of 9 weeks) during pharmacological counseling.
  Data from medical records for 5 years follow-up will be used to investigate adherence to recommendations during pharmacologic counseling and in a long term perspective.
Prediction of long-term prognosis of depressive symptom profiles | 5 years follow-up from baseline visit
  Data on clinical outcome over 5 years follow-up for depressive symptom profiles with specific focus on anhedonic symtom profile derived from the Comprehensive Psychopatholocial Rating Scale (CPRS) and depression characteristics.
Course of disease related to dopamine D3 receptor and other biomarkers | 5 years follow-up from baseline visit
  The relationship between the course of depressive disorder and biomarkers including dopamine D3 receptor, other biomarkers of dopaminergic function, inflammation and other types of biomarkers

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Psychiatry Reserach Unit, Lund
  - Research Unit, Office of Psychiatricy, habilitation and technical aid, Lund

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Asp M, Lindqvist D, Fernstrom J, Ambrus L, Tuninger E, Reis M, Westrin A. Recognition of personality disorder and anxiety disorder comorbidity in patients treated for depression in secondary psychiatric care. PLoS One. 2020 Jan 2;15(1):e0227364. doi: 10.1371/journal.pone.0227364. eCollection 2020. PMID 31895938
- [Background] Asp M, Ambrus L, Reis M, Manninen S, Fernstrom J, Lindqvist D, Westrin A. Differences in antipsychotic treatment between depressive patients with and without a suicide attempt. Compr Psychiatry. 2021 Aug;109:152264. doi: 10.1016/j.comppsych.2021.152264. Epub 2021 Jul 8. PMID 34271258
- [Background] Soderberg Veiback G, Malmgren L, Asp M, Ventorp F, Suneson K, Grudet C, Westrin A, Lindqvist D. Inflammatory depression is associated with selective glomerular hypofiltration. J Affect Disord. 2024 Jul 1;356:80-87. doi: 10.1016/j.jad.2024.04.007. Epub 2024 Apr 2. PMID 38574872
- [Background] Suneson K, Grudet C, Ventorp F, Malm J, Asp M, Westrin A, Lindqvist D. An inflamed subtype of difficult-to-treat depression. Prog Neuropsychopharmacol Biol Psychiatry. 2023 Jul 13;125:110763. doi: 10.1016/j.pnpbp.2023.110763. Epub 2023 Apr 8. PMID 37037323
- [Background] Grudet C, Wolkowitz OM, Mellon SH, Malm J, Reus VI, Brundin L, Nier BM, Dhabhar FS, Hough CM, Westrin A, Lindqvist D. Vitamin D and inflammation in major depressive disorder. J Affect Disord. 2020 Apr 15;267:33-41. doi: 10.1016/j.jad.2020.01.168. Epub 2020 Jan 29. PMID 32063570
- [Background] Fernstrom J, Ohlsson L, Asp M, Lavant E, Holck A, Grudet C, Westrin A, Lindqvist D. Plasma circulating cell-free mitochondrial DNA in depressive disorders. PLoS One. 2021 Nov 4;16(11):e0259591. doi: 10.1371/journal.pone.0259591. eCollection 2021. PMID 34735532
- [Background] Holck A, Asp M, Green H, Westrin A, Reis M. CYP2D6 Genotyping and Inhibition as Predictors of Adverse Drug Reactions in Depressive Disorders. J Clin Psychiatry. 2024 Jan 17;85(1):23m14937. doi: 10.4088/JCP.23m14937. PMID 38236047
- [Background] Ambrus L, Sunnqvist C, Asp M, Westling S, Westrin A. Coping and suicide risk in high risk psychiatric patients. J Ment Health. 2020 Feb;29(1):27-32. doi: 10.1080/09638237.2017.1417547. Epub 2017 Dec 20. PMID 29260914